CLINICAL TRIAL: NCT00364624
Title: Adrenal Cortical Function in Patients With Newly Diagnosed Lung Cancer
Brief Title: Adrenal Function in Patients With Newly Diagnosed Lung Cancer
Status: Completed | Type: Observational
Sponsor: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Dr. W C Yu, Consultant Physician, Princess Margaret Hospital, Hong Kong
Other Study IDs: KW/FR/06-008
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Lung Cancer; Adrenal Insufficiency
Keywords: lung cancer; adrenal insufficiency
MeSH Terms: conditions — Lung Neoplasms; Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with newly diagnosed lung cancer may have hypofunction of the adrenal cortex either from tumour metastasis or other mechanisms. Since lung cancer patient may have to undergo stressful investigation and treatments, undetected hypofunction of the adrenal cortex may be hazardous. Knowledge of the size of the problem may help determine whether routine check is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary lung cancer
* Newly diagnosed
* No specific treatment given
* No active infection in the previous week
* No general anesthesia in the previous week

Exclusion Criteria:

* Known adrenal disease
* Receiving exogenous systemic corticosteroids
* Concomitant illness known to affect adrenal function. e.g. active TB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed, histologically confirmed primary lung cancer
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wai C YU, MBBS, Principal Investigator — Princess Margaret Hospital, Hong Kong
Locations (1):
- Department of Medicine, Princess Margaret Hospital, Kowloon, Hong Kong SAR, China